CLINICAL TRIAL: NCT06613737
Title: An Exploratory Study to Establish the Dose, Safety and Pathogenicity of a New Influenza A H3N2 Challenge Strain in Healthy Participants 18 to 55 Years of Age
Brief Title: Dose, Safety, and Pathogenicity of a New Influenza A H3N2 Challenge Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HRD-vCS-006
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Influenza A H3N2
Keywords: Influenza; Flu; H3N2; Human Challenge Trial
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose 1 (Experimental): Medium dose, expected to be approximately 10^5.5 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Interventions: Other: Influenza A H3N2 virus dose arm 1
- Dose 2 (Experimental): High dose, expected to be approximately 10^4 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Interventions: Other: Influenza A H3N2 virus dose arm 2
- Dose 3 (Experimental): Optional: TBD, depending on outcome of Part A
  Interventions: Other: Influenza A H3N2 virus dose arm 3

INTERVENTIONS:
Other: Influenza A H3N2 virus dose arm 1 — Medium dose, approximately 10^4.5 TCID50/mL
  Arms: Dose 1
Other: Influenza A H3N2 virus dose arm 2 — High dose, approximately 10^5.5 TCID50/mL
  Arms: Dose 2
Other: Influenza A H3N2 virus dose arm 3 — TBD, depending on outcome of Part A
  Arms: Dose 3

SUMMARY:
An Exploratory Study to Establish the Dose, Safety and Pathogenicity of a New Influenza A H3N2 Challenge Strain in Healthy Participants 18 to 55 Years of Age

In Part A, up to 40 participants will be randomly allocated to one of two groups to be given one of two virus doses (Virus Dose 1 or Virus Dose 2).

Based on the outcome of Part A, participants in Part B, may be given Virus Dose 1, Virus Dose 2, or another virus dose (e.g., Virus Dose 3)

DETAILED DESCRIPTION:
This is an exploratory study of an influenza A/England/7763/2022 H3N2 challenge strain, to determine the optimum safe infectious titer of challenge agent, in healthy participants 18 to 55 years of age.

A total of up to 80 participants may be given the influenza A/England/7763/2022 H3N2 challenge agent. Each participant will remain in the study for approximately 4 months from screening to the last clinic visit.

The study will consist of 2 parts, in Part A of the study, up to 40 participants will be randomly allocated to one of two groups to be given one of two virus doses (Virus Dose 1 or Virus Dose 2). Based on the outcome of Part A, additional participants may be enrolled into the optional Part B of the study and may be given Virus Dose 1, Virus Dose 2, and/or another virus dose (e.g., Virus Dose 3)

The study is divided into three phases:

1. Screening phase: Screening will occur between Day -90 to Day -2/-1.
2. Quarantine phase: Participants will stay in the quarantine unit for approximately 8 days (from Day -2/-1 to Day 8).

   One or two days prior to the day of inoculation with the challenge virus, participants will be admitted to quarantine where their eligibility will be reassessed. If participants remain eligible for the study, they will receive the challenge virus on Day 0. Participants will undergo a range of clinical assessments and safety monitoring for the entirety of their stay in quarantine. Participants will be discharged from the quarantine unit on Day 8 (or may remain longer at the principal investigator's discretion).
3. Outpatient phase: Following the conclusion of the quarantine phase, participants will attend a Follow-Up visit, approximately 28 days after they received the study virus. Their symptoms will be reassessed, and a complete safety examination performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult male or female aged between 18 and 55 years
* A total body weight ≥50 kg and body mass index (BMI) ≥18 kg/m2 and ≤35kg/m2.
* In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety.
* Documented medical history
* Adherence to contraception requirements
* Serosuitable for the challenge virus

Exclusion Criteria:

* History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit.
* Any history or evidence of any clinically significant or currently active disease.
* Any participants who have smoked ≥10 pack years at any time.
* Female participants who are breastfeeding, or have been pregnant within 6 months prior to the study, or have a positive pregnancy test at any point during screening or prior to inoculation.
* Any history of anaphylaxis and/or a any history of severe allergic reaction.
* Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
* Lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction.
* Significant abnormality of the nose, includes loss of or alterations in smell or taste, nasal polyps, epistaxis, nasal or sinus surgery.
* Recent vaccinations or intention to receive vaccination before the Day 28 follow up visit.
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned inoculation or planned during the 3 months after the final visit.
* Recent receipt of investigational drugs or challenge viruses.
* Use or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows.
* Positive drugs of abuse test, recent history or presence of alcohol addiction, excessive consumption of xanthine containing substances or a presence of significant signs and symptoms of nicotine withdrawal on first study visit.
* A forced expiratory volume in 1 second (FEV1) <80%.
* Positive HIV, hepatitis B virus, or hepatitis C virus test.
* Presence of fever, defined as participant presenting with a temperature reading of ≥37.9°C on Day -2/-1 and/or pre-inoculation on Day 0.
* Those employed or immediate relatives of those employed at hVIVO or the sponsor.
* Any other reason, in the opinion of the investigator deems the participant unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events related to the viral challenge | Day 0 to Day 28
  Occurrence of adverse events (AEs) related to the viral challenge from viral challenge (Day 0) to the Day 28 follow-up visit.
Occurrence of serious adverse events related to the viral challenge | Day 0 to Day 28
  Occurrence of serious adverse events (SAEs) related to the viral challenge from viral challenge (Day 0) to the Day 28 follow-up visit.
Induces laboratory-confirmed infection in ≥40% of inoculated participants | Day 1 to Day 8
  Quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR)-confirmed influenza infection, defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (reported over 4 planned consecutive assessments within 48 hours), from Day 1 pm to planned discharge from quarantine (Day 8 am).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lima, MD-PhD, Principal Investigator — hVIVO Services Ltd.
Locations (1):
- hVIVO Services Ltd, 40 Bank Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No